CLINICAL TRIAL: NCT00018759
Title: Treatment Effects on Platelet Calcium in Hypertensive and Depressed Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: SmithKline Beecham (Industry)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHBS-023-00S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Depression; Hypertension
Keywords: Serotonin, Hypertension, Depression
MeSH Terms: conditions — Depression; Hypertension | interventions — Paroxetine

INTERVENTIONS:
Drug: paroxetine
Behavioral: ongoing psychological screening

SUMMARY:
This study aims to determine if treatment with an SSRI antidepressant medication, paroxetine, is associated with cellular calcium response to serotonin, platelet serotonin receptors, and improvement in mood in depressed patients with or without hypertension. It is hypothesized that platelets of hypertensive patients with depressive symptomatology with be hyper-responsive to serotonin. Additionally, treatment with an SSRI antidepressant is expected to produce a down-regulation of the serotonin receptor with an associated reduction in platelet cytosolic calcium response as well as improved mood.

ELIGIBILITY:
Subjects for all study groups will be male and between the ages of 25 and 65

Hypertension & Depression Group: Hypertension controlled with an ACE-inhibitor anti-hypertensive; no co-morbid medical conditions known to influence psychological functioning or platelet calcium responses including uncontrolled diabetes, MI or CVA within 6 months of enrollment, secondary hypertension; depression as diagnosed by structured interview and HDRS score of 18; no active participation in another clinical trial; no current suicidal/ homicidal ideation

Hypertension Group: Hypertension controlled with an ACE-inhibitor anti-hypertensive; no co-morbid medical conditions known to influence psychological functioning or platelet calcium responses including uncontrolled diabetes, MI or CVA within 6 months of enrollment, secondary hypertension; no active participation in another clinical trial; no current suicidal/ homicidal ideation

Depression Group: No co-morbid medical conditions known to influence psychological functioning or platelet calcium responses including uncontrolled diabetes, MI or CVA within 6 months of enrollment, secondary hypertension; depression as diagnosed by structured interview and HDRS score of 18; no active participation in another clinical trial; no current suicidal/ homicidal ideation

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Study Completion 2003-10

CONTACTS AND LOCATIONS:
Locations (1):
- Edward Hines Jr. Hospital, Hines, Illinois, United States